CLINICAL TRIAL: NCT05392881
Title: University of Kansas Medical Center Interstitial Lung Disease Research Unit (ILDRU) Biobank
Brief Title: Interstitial Lung Disease Research Unit Biobank
Acronym: ILDRU
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Scott Matson, Assistant Professor of Medicine, University of Kansas Medical Center
Other Study IDs: STUDY00144558
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Interstitial Lung Disease; Sarcoidosis; Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Hypersensitivity Pneumonitis
Keywords: Interstitial Lung Disease; Sarcoidosis; Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Hypersensitivity Pneumonitis
MeSH Terms: conditions — Lung Diseases, Interstitial; Sarcoidosis; Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Alveolitis, Extrinsic Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Establish a interstitial lung disease (ILD) registry and biorepository to lead towards a further understanding of the disease.

DETAILED DESCRIPTION:
The University of Kansas ILD and Rare Lung Disease clinic sees hundreds of new patients per year. The investigators would like to leverage this resource to develop an Interstitial Lung Disease Research Unit (ILDRU) repository and database to help develop new methods for early diagnosis, uncover underlying genetic and environmental risk factors, as well as potential treatment targets in the broad range of interstitial lung diseases and rare lung diseases (RLD).

ELIGIBILITY:
Inclusion Criteria:

1. The participant is a patient at TUKHS or has agreed to participate in a study approved by the KUMC Human Research Protection Program (HRPP)
2. The participant is being followed for the presence of autoimmune disease, ILD or other rare lung diseases at TUKHS.
3. The participant is ≥ 18 years of age.
4. The participant has signed an approved consent for this study (living patients only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ILD, RLD and subjects at risk for ILD
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2031-08-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Collect clinically obtained data for patients with ILD, RLD and risk for ILD/RLD to support research. | Enrollment to Year 10
Establish a collection of biological samples from patients with ILD, RLD and subjects at risk for ILD. | Enrollment to Year 10
Correlate biological samples with individual longitudinal clinical data. | Enrollment to Year 10
Provide biological samples to researchers performing studies in ILD and RLD. | Enrollment to Year 10
Collect historical data and imaging from deceased patients with ILD. | Enrollment to Year 10

CONTACTS AND LOCATIONS:
Overall Officials: Scott Matson, M.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact Kimberly Lovell to discuss accessing IPD